CLINICAL TRIAL: NCT07243626
Title: Efficacy and Safety of Envafolimab Combined With Doxorubicin and Ifosfamide as First-line Treatment for Advanced Soft Tissue Sarcoma
Brief Title: Efficacy and Safety of Envafolimab Plus Doxorubicin and Ifosfamide for Advanced Soft Tissue Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR2023375
Record Dates: First submitted 2025-09-24; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention (Experimental): Eligible patients with soft tissue sarcoma were enrolled and treated with Envafolimab 300 mg/dose subcutaneously every 3 weeks on day 1. The AI regimen consisted of liposomal doxorubicin 35 mg/m² on day 1 and intravenous infusion of IFO 2.5 mg/m² on days 1-3, every 3 weeks. Efficacy and safety were assessed approximately every 6 weeks (42 ± 7 days). Patients with disease control (CR+PR+SD) and tolerable adverse reactions could continue treatment until disease progression, unacceptable toxicity, or discontinuation at the investigator's discretion.
  Interventions: Drug: Envafolimab combined with an AI regimen (doxorubicin and ifosfamide)

INTERVENTIONS:
Drug: Envafolimab combined with an AI regimen (doxorubicin and ifosfamide) — Envafolimab combined with an AI regimen: liposomal doxorubicin 35 mg/m² on day 1; IFO 2.5 mg/m² on days 1-3, intravenous infusion, every 3 weeks.

SUMMARY:
Soft tissue sarcoma (STS) is a rare, highly heterogeneous malignancy with a poor prognosis. The standard first-line treatment for advanced patients is anthracyclines (doxorubicin, A) combined with ifosfamide (I, AI regimen), but the efficacy is limited, and some subtypes do not respond well. Immune checkpoint inhibitors (ICI) have shown potential in specific STS subtypes. Anthracyclines can induce immunogenic cell death and upregulate PD-L1, providing a theoretical basis for combined immunotherapy. Previous studies have shown that ICI combined with chemotherapy (such as pembrolizumab + doxorubicin) is more effective than chemotherapy alone. Envolizumab is the world's first subcutaneously injected PD-L1 single-domain antibody-Fc fusion protein, with significant advantages: (1) small molecular weight (~80kDa) and strong tissue penetration; (2) high stability and can be stored at room temperature; (3) convenient subcutaneous injection and good tolerability (Phase II study of MSI-H/dMMR solid tumors ORR 42.7%, grade 3-4 TEAE 15.5%). In 2022, the FDA granted orphan drug designation for the treatment of STS.

This study aims to evaluate the efficacy (ORR, PFS, OS, etc.) and safety of Envolizumab combined with an AI regimen (doxorubicin + ifosfamide) as a first-line treatment for advanced STS.

DETAILED DESCRIPTION:
Soft tissue sarcoma (STS) encompasses a diverse group of rare, high-grade malignancies originating from mesenchymal tissues, exhibiting significant heterogeneity in histology, molecular characteristics, and clinical behavior. The prognosis for advanced or metastatic STS remains generally poor, underscoring the urgent need for more effective therapeutic strategies. Currently, the standard first-line treatment for advanced STS involves chemotherapy regimens comprising anthracyclines, primarily doxorubicin, often combined with ifosfamide (the AI regimen). While these regimens can induce tumor responses, their overall efficacy is limited, with modest response rates and survival benefits. Moreover, certain STS subtypes demonstrate resistance to conventional chemotherapy, highlighting the necessity for novel and combination treatment approaches.

Recent advances in immunotherapy, particularly immune checkpoint inhibitors (ICIs) targeting PD-1/PD-L1 pathways, have opened new avenues for treating specific STS subtypes. Evidence suggests that anthracyclines, such as doxorubicin, can induce immunogenic cell death, enhance tumor antigen presentation, and upregulate PD-L1 expression, creating a compelling rationale for combining chemotherapy with immunotherapy. Indeed, clinical studies have demonstrated that combining ICIs like pembrolizumab with chemotherapy regimens can improve objective response rates (ORR), progression-free survival (PFS), and overall survival (OS) compared to chemotherapy alone in certain patient populations.

Envolizumab represents a groundbreaking development in the realm of immunotherapeutics. As the world's first subcutaneously injectable PD-L1 single-domain antibody-Fc fusion protein, it boasts several distinct advantages: a small molecular weight (~80 kDa) that ensures superior tissue penetration, high stability with room temperature storage capability, and a convenient subcutaneous administration route that enhances patient tolerability and adherence. Phase II clinical data have demonstrated promising anti-tumor activity in MSI-H/dMMR solid tumors, with an ORR of 42.7%, and an acceptable safety profile, with grade 3-4 treatment-emergent adverse events (TEAEs) in only 15.5% of patients. Notably, in 2022, the FDA granted orphan drug designation to Envolizumab for the treatment of STS, highlighting its potential as a novel therapeutic option.

This study aims to systematically evaluate the efficacy and safety of combining Envolizumab with the AI chemotherapy regimen as a first-line treatment for patients with advanced STS. The primary endpoint will focus on the overall response rate (ORR), with secondary endpoints including disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and safety profile assessments. The study hypothesizes that this combination could synergistically enhance anti-tumor immune responses, improve clinical outcomes, and offer a more tolerable treatment option for patients with advanced STS. The findings could potentially establish a new standard of care and provide critical insights into the integration of immunotherapy and chemotherapy in the management of this challenging malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed advanced soft tissue sarcoma with at least one measurable lesion.
2. No previous systemic treatment.
3. ≥18 years old; ECOG score: 0 or 1; expected survival time more than 3 months;
4. Major organ function within 7 days before treatment, meeting the following criteria:

(1) Routine blood test criteria (without blood transfusion within 14 days):

* Hemoglobin (HB) ≥90g/L; ② Absolute neutrophil count (ANC) ≥1.5×109/L; ③ Platelet count (PLT) ≥80×109/L. (2) Biochemical examinations must meet the following criteria: ① Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); ② Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5 ULN. If liver metastasis is present, ALT and AST ≤ 5 ULN; ③ Serum creatinine (Cr) ≤ 1.5 ULN or creatinine clearance (CCr) ≥ 60ml/min; (3) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%). 5. Women of childbearing age must agree to use contraceptive measures (such as intrauterine devices, birth control pills or condoms) during the study and within 6 months after the study; serum or urine pregnancy tests must be negative within 7 days before study enrollment, and the patients must not be breastfeeding; men must agree to use contraceptive measures during the study and within 6 months after the study.

Exclusion Criteria:

1. Chondrosarcoma (CS), osteosarcoma (OS), Ewing's sarcoma, dermatofibrosarcoma protuberans (DFSP), and gastrointestinal stromal sarcoma (GIST) are excluded;
2. Pregnant or lactating women, or women of childbearing potential who are not using contraceptive measures;
3. Current severe, uncontrolled acute infection; or purulent or chronic infection with a persistent wound;
4. Presence of a second primary tumor (excluding basal cell carcinoma of the skin);
5. Participation in other drug clinical trials within 4 weeks;
6. Presence of severe heart disease, including congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina, myocardial infarction, severe valvular heart disease, and refractory hypertension;
7. Suffering from uncontrolled neurological, psychiatric, or mental disorders, poor compliance, and inability to match the medication. Patients with uncontrolled primary brain tumors or central nervous system metastases and significant intracranial hypertension or neuropsychiatric symptoms are excluded.
8. Evidence of a hereditary bleeding diathesis or coagulopathy.
9. A history of severe allergic/anaphylactic reactions to humanized antibodies.
10. Diagnosed with immunodeficiency or receiving systemic glucocorticoids or any other form of immunosuppressive therapy within 14 days prior to the first dose of the study drug. Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are permitted.
11. Subjects with active, known, or suspected autoimmune diseases (e.g., interstitial pneumonitis, colitis, hepatitis, hypophysitis, vasculitis, nephritis, including but not limited to these diseases or syndromes) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Efficcy-Objective response rate | From enrollment to the end of treatment at 8 weeks
  Objective response rate(ORR) =CR+PR

SECONDARY OUTCOMES:
Efficcy-Disease control rate | From enrollment to the end of treatment at 8 weeks
  DCR=CR+PR+SD
Efficcy-Progression-free survival | From enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS
Efficcy-overall survival | From enrollment until the date of death from any cause, assessed up to 60 months
  OS
adverse events-safety | From enrollment to the end of treatment at 8 weeks
  adverse events

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: 2025.8.3-2026-9.1